CLINICAL TRIAL: NCT00295230
Title: The Effects of Volume Guarantee Combined With Pressure Supported Ventilation (PSV+VG) Versus Synchronized Intermittent Mandatory Ventilation (SIMV+VG) in Very Low Birth Weight Infants
Brief Title: Effects of Volume Guarantee With Pressure Supported vs. Synchronized Intermittent Mandatory Ventilation in VLBW Infants
Status: Suspended | Type: Observational
Why Stopped: suboptimal enrollment after 18 months.
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Collaborators: Windtree Therapeutics (Industry)
Other Study IDs: 0512098
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2007-11-07 (Estimated); Status verified 2007-11

CONDITIONS: Respiratory Distress Syndrome
Keywords: respiratory distress syndrome; very low birth weight infant; mechanical ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

INTERVENTIONS:
Procedure: PSV+VG mode versus SIMV+VG mode — fully assisted mechanical ventilation versus assistance on only a select number of breaths

SUMMARY:
Studies in preterm infants have shown that adding volume guarantee (VG) to synchronized modes of ventilation is not only feasible but also advantageous for providing more constant and desirable mechanical breath size. This ideally minimizes ventilator-induced lung injury due to barotrauma and volutrauma. To date, only one recent study has investigated the relative advantages of combining VG with different modes of synchronized mechanical ventilation in clinically stable, preterm infants that were mechanically ventilated at an average age of one month. We aim to further evaluate the effects of PSV+VG versus SIMV+VG ventilation in very low birth weight infants within the first three to five days of life. Our hypothesis is that in very low birth weight infants requiring mechanical ventilation in the first three to five days of life, PSV+VG will allow for more stable physiologic and ventilatory parameters compared to SIMV+VG. The primary endpoints are a reduction in respiratory rate and average mean airway pressure in the PSV+VG group compared to the SIMV+VG group.

DETAILED DESCRIPTION:
After informed consent is obtained, each patient will be started on the study between 72 to 96 hours of age. Each infant will be assigned via block randomization to an initial ventilation mode (PSV+VG or SIMV+VG). Mechanical ventilation will be provided using the Dräeger Babylog 8000Ò. Once on study, infants will receive each ventilation mode (PSV+VG and SIMV+VG) twice, administered in alternating ninety minute blocks. Ventilator management in each mode will be standardized as follows: ventilator rate of 30 breaths per minute, volume guarantee of 4-6 cc/kg, inspiratory time of 0.3-0.35 seconds, and positive end-expiratory pressure of 5-7 cmH2O. Peak inspiratory pressure (PIP) will be set at 15-20% above the PIP needed to achieve the set tidal volume. FiO2 will be maintained to keep oxygen saturation in the range of 85-96%. The FiO2 will only be adjusted if the infant's oxygen saturation is persistently outside of the target range. End tidal carbon dioxide levels will be obtained at two times (30 minutes and 90 minutes) during each study block.

No laboratory tests will be obtained for this study. However, blood gases may be obtained by the NICU care team during the study per their daily care plan, and subsequent ventilator changes may be made by the NICU care team if necessary to correct an undesired blood gas value.

All data will be obtained using the pre-existing equipment in place to care for the patient prior to this study. This equipment includes the mechanical ventilator, endotracheal tube, cardio-respiratory monitor, and blood pressure monitor.

The key measurements during this study are ventilator variables and physiologic vital signs. Ventilator variables include respiratory rate, actual PIP, mean airway pressure, FiO2, expiratory tidal volume, minute ventilation, and actual I-time. Vital signs include heart rate, oxygen saturation, and blood pressure. Ventilator variables will be continuously downloaded from the Dräeger Babylog 8000Ò using BabyviewÒ software. Heart rate and oxygen saturation data will be downloaded from the MassimoÒ pulse oximeter. Blood pressure measurements will be documented every ten minutes if the infant has an umbilical artery catheter (UAC) or percutaneous arterial line (PAL) in place. If the infant does not have an UAC or PAL in place prior to the study, blood pressure measurements will be obtained every thirty minutes via manual blood pressure cuff.

ELIGIBILITY:
Inclusion Criteria:

* Infants will be recruited based on the following criteria: weight ≤1500 grams and need for mechanical ventilation at 72 - 120 hours of age. Recruitment will continue until 16 patients have completed the study

Exclusion Criteria:

* Exclusion criteria include significant endotracheal tube leak (>30% leak does not allow for accurate measurement of ventilator data), use of narcotic drip medication, use of paralytic medication, use of inhaled nitric oxide, fraction of inspired oxygen (FiO2) >70% at the time of enrollment, or significant congenital defects of any organ system (e.g. cardiac, respiratory, CNS).

Ages: 72 Hours to 120 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: premature infants weighing </= 1500 grams and needing mechanical ventilation at 72-120 hours of age.
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2006-02; Study Completion 2007-09 (Estimated)

PRIMARY OUTCOMES:
Respiratory rate | 6hr

SECONDARY OUTCOMES:
Ventilator variables | 6hr
Vital signs | 6hr

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mammel, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Cheema IU, Ahluwalia JS. Feasibility of tidal volume-guided ventilation in newborn infants: a randomized, crossover trial using the volume guarantee modality. Pediatrics. 2001 Jun;107(6):1323-8. doi: 10.1542/peds.107.6.1323. PMID 11389251
- [Background] Herrera CM, Gerhardt T, Claure N, Everett R, Musante G, Thomas C, Bancalari E. Effects of volume-guaranteed synchronized intermittent mandatory ventilation in preterm infants recovering from respiratory failure. Pediatrics. 2002 Sep;110(3):529-33. doi: 10.1542/peds.110.3.529. PMID 12205255
- [Background] Keszler M, Abubakar K. Volume guarantee: stability of tidal volume and incidence of hypocarbia. Pediatr Pulmonol. 2004 Sep;38(3):240-5. doi: 10.1002/ppul.20063. PMID 15274104
- [Background] Mrozek JD, Bendel-Stenzel EM, Meyers PA, Bing DR, Connett JE, Mammel MC. Randomized controlled trial of volume-targeted synchronized ventilation and conventional intermittent mandatory ventilation following initial exogenous surfactant therapy. Pediatr Pulmonol. 2000 Jan;29(1):11-8. doi: 10.1002/(sici)1099-0496(200001)29:13.0.co;2-5. PMID 10613781
- [Background] Abubakar K, Keszler M. Effect of volume guarantee combined with assist/control vs synchronized intermittent mandatory ventilation. J Perinatol. 2005 Oct;25(10):638-42. doi: 10.1038/sj.jp.7211370. PMID 16094389